CLINICAL TRIAL: NCT03324113
Title: A Phase I Study to Evaluate Safety and Pharmacokinetics of SAR408701 Administered Intravenously as Monotherapy in Japanese Patients With Advanced Malignant Solid Tumors
Brief Title: Evaluation of SAR408701 in Japanese Patients With Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TCD15054; U1111-1191-5464 (Registry Identifier: ICTRP); TCD15054 (Other: Sanofi Identifier)
Record Dates: First submitted 2017-10-06; First posted 2017-10-27 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — tusamitamab ravtansine; Dexamethasone; Naphazoline; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SAR408701 Monotherapy (Experimental): SAR408701 Dose escalation administered as a single agent intravenously, on Day 1 and once every two weeks, to patients with malignant solid tumors
  Interventions: Drug: SAR408701; Drug: dexamethasone; Drug: naphazoline; Drug: diphenhydramine

INTERVENTIONS:
Drug: SAR408701 — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Other Names: Tusamitamab ravtansine
Drug: dexamethasone — Pharmaceutical form: solution for eye drop
  Route of administration: eye drop
  Other Names: Santeson ophthalmic solution
Drug: naphazoline — Pharmaceutical form: solution for eye drop
  Route of administration: eye drop
  Other Names: Clearine
Drug: diphenhydramine — Pharmaceutical form: tablet
  Route of administration: oral
  Other Names: Restamin Kowa

SUMMARY:
Primary Objective:

* To evaluate tolerability and safety of SAR408701 when administered as a single agent according to the investigational medicinal product (IMP) related dose limiting toxicities (DLTs) to determine the recommended dose (RD) of SAR408701 in Japanese patients with advanced malignant solid tumors.

Secondary Objectives:

* To characterize the overall safety profile of SAR408701 monotherapy.
* To characterize the pharmacokinetic (PK) profile of SAR408701 and its metabolites.
* To evaluate the pharmacodynamic (PDy) effect of SAR408701 on levels of circulating carcinoembryonic antigen-related cell adhesion molecule 5 (CEACAM5) for main dose escalation part.
* To assess preliminary efficacy according to Response Evaluation Criteria in Solid Tumor (RECIST) 1.1 criteria and other indicators of antitumor activity.
* To assess the potential immunogenicity of SAR408701.

DETAILED DESCRIPTION:
The study duration per participant will include a period to assess eligibility (screening period) of up to approximately 4 weeks (28 days), a treatment period and an End-of-Treatment (EOT) visit around 30 days after the last administration of IMP, and at least one follow-up (FU) visit after the EOT visit.

ELIGIBILITY:
Inclusion criteria:

* Locally advanced or metastatic solid malignant tumor disease for which, in the judgement of the investigator, no standard alternative therapy is available.
* Inclusion is likely to be expressing CEACAM5.
* At least 6 x 5 μm slides from formalin-fixed paraffin-embedded (FFPE) archival tissue should be available for retrospective central evaluation of CEACAM5 expression.
* Patient understands and has signed the Written Informed Consent form and is willing and able to comply with the requirements of the trial.

Exclusion criteria:

* Patient less than 20 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≥2.
* Life expectancy <12 weeks.
* Known or symptomatic brain metastasis (other than totally resected or previously irradiated and non-progressive/relapsing) or lepto-meningeal carcinomatosis.
* Female patients of childbearing potential and male patients with female partners of childbearing potential who do not agree to use accepted and effective method of contraception during the study treatment period and for 6 months following discontinuation of IMP.
* Significant concomitant illnesses, including all severe medical conditions which, in the opinion of the Investigator or Sponsor, would impair the patient's participation in the study or interpretation of the results.
* Prior therapy targeting CEACAM5.
* Prior maytansinoid treatments (maytansinoid derivative 1 [DM1] or maytansinoid derivative 4 [DM4] antibody drug conjugates).
* Previous history and or unresolved corneal disorders.
* Medical conditions requiring concomitant administration of medications with narrow therapeutic window, metabolized by cytochrome P450 (CYP) and for which a dose reduction cannot be considered.
* Medical conditions requiring concomitant administration of strong CYP3A inhibitor, unless it can be discontinued at least 2 weeks before first administration of SAR408701.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-12-26 (Actual)

PRIMARY OUTCOMES:
IMP-related dose limiting toxicities (DLT) | 4 weeks, Dose escalation q3w part: 3 weeks
  IMP-related DLTs are defined as adverse events (AE) related to the IMPs in absence of clear evidence to the contrary, after validation by the Study Committee, and if not related to a disease progression, graded using National Cancer Institute common Toxicity Criteria (NCI-CTC) scale v4.03

SECONDARY OUTCOMES:
Treatment emergent adverse events | Up to an average of 9 months
  Overall safety profile characterized in terms of the type, frequency, severity, seriousness, and relationship to study therapy of any AEs based on standard and systematic assessment including physical findings, laboratory tests or other investigations
Maximum observed concentration (Cmax) of SAR408701 | Main dose-escalation part: Cycle 1 and Cycle 4 (each cycle is 14 days); Dose-escalation bis part with loading dose: Cycle 1 (Cycle 1 is 14 days), Dose-escalation q3w part: Cycle 1 and Cycle2 day 1 (Cycle 1 is 21 days)
  Cmax for SAR408701 will be assessed after single and repeat doses, as relevant
Cmax of DM4 and Me-DM4 | Main dose-escalation part: Cycle 1 and Cycle 4 (each cycle is 14 days); Dose-escalation bis part with loading dose: Cycle 1 (Cycle 1 is 14 days), Dose-escalation q3w part: Cycle 1 and Cycle2 day 1 (Cycle 1 is 21 days)
  Cmax for DM4 and Me-DM4 will be assessed after single and repeat doses, as relevant
Time to reach maximum concentration (Tmax) of SAR408701 | Main dose-escalation part: Cycle 1 and Cycle 4 (each cycle is 14 days); Dose-escalation bis part with loading dose: Cycle 1 (Cycle 1 is 14 days), Dose-escalation q3w part: Cycle 1 and Cycle2 day 1 (Cycle 1 is 21 days)
  Tmax for SAR408701 will be assessed after single and repeat doses, as relevant
Tmax of DM4 and Me-DM4 | Main dose-escalation part: Cycle 1 and Cycle 4 (each cycle is 14 days); Dose-escalation bis part with loading dose: Cycle 1 (Cycle 1 is 14 days), Dose-escalation q3w part: Cycle 1 and Cycle2 day 1 (Cycle 1 is 21 days)
  Tmax for DM4 and Me-DM4 will be assessed after single and repeat doses, as relevant
Area under the concentration-time curve (AUC) of SAR408701 | Main dose-escalation part: Cycle 1 and Cycle 4 (each cycle is 14 days); Dose-escalation bis part with loading dose: Cycle 1 (Cycle 1 is 14 days), Dose-escalation q3w part: Cycle 1 and Cycle2 day 1 (Cycle 1 is 21 days)
  AUC of SAR408701 from time zero extrapolated to infinity
AUC of DM4 and Me-DM4 | Main dose-escalation part: Cycle 1 and Cycle 4 (each cycle is 14 days); Dose-escalation bis part with loading dose: Cycle 1 (Cycle 1 is 14 days), Dose-escalation q3w part: Cycle 1 and Cycle2 day 1 (Cycle 1 is 21 days)
  AUC of DM4 and Me-DM4 from time zero extrapolated to infinity
Assessment of PDy effect | Up to an average of 10 months
  Assessment of plasma CEACAM5 levels in main dose-escalation part
Assessment of anti-tumor activity | Up to an average of 10 months
  Assessment of tumor response using standard imaging, as defined by RECIST 1.1 criteria
Detection of anti-SAR408701 antibody | Up to an average of 10 months
  Immunogenicity evaluation for anti-SAR408701 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- Japan (3):
  - Investigational Site Number : 3920002, Nagoya, Aichi-ken
  - Investigational Site Number : 3920003, Kashiwa-shi, Chiba
  - Investigational Site Number : 3920001, Sunto-gun, Shizuoka

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Muro K, Yamazaki K, Kadowaki S, Mishima S, Kawakami T, Tanaka T, Tada K, Fagniez N, Ohshima S, Yoshino T. Phase 1 study evaluating safety and pharmacokinetics of tusamitamab ravtansine monotherapy in Japanese patients with advanced malignant solid tumors. Int J Clin Oncol. 2025 Aug;30(8):1522-1536. doi: 10.1007/s10147-025-02784-4. Epub 2025 May 25. PMID 40413667